CLINICAL TRIAL: NCT06337019
Title: Multicentric, Observational, Longitudinal Study for the Evaluation of Nutritional Management Implications in Newly Diagnosed Italian Cancer Patients: The Italian Registry of Malnutrition in Oncology (IRMO)
Brief Title: The Italian Registry of Malnutrition in Oncology
Acronym: IRMO
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Sponsor
Other Study IDs: IRMO
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Cancer Metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort observational: Overall study cohort
  Interventions: Other: Cohort observational

INTERVENTIONS:
Other: Cohort observational — Cohort observational

SUMMARY:
The aim of the Italian Registry of Malnutrition in Oncology (IRMO) is to set up a digital register of newly diagnosed or treated oncologic patients to monitor their nutritional status, early identify malnutrition and investigate the implications of nutritional support management. In particular, this project aims to establish a prospective cohort of cancer patients in order to investigate the effects of nutritional status and management on overall survival (OS) and progression free survival (PFS), and analyse the effects of the nutritional management and support on patients' symptoms and QoL.

DETAILED DESCRIPTION:
This is a multicentric longitudinal observational study on a cohort of newly diagnosed cancer patients, candidate for active treatment. In Italy, no reliable data are still available with regards to the actual implementation of adequate nutritional support management in cancer patients; only "real-world" data collected by administrative databases are available in the context of nutrition in oncology, and this somehow limits the possibility to interpret the evidence from a clinical point of view. Hence, the purpose of the intestigators is to collect "real world" clinical data on malnutrition in oncology at the national level, in order to strengthen the evidence and concretely improve nutritional care practices in oncology.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years;
* New diagnosis of the following cancers: head and neck, oesophagus/stomach, colorectal, hepato-biliary, pancreatic, lung, prostate, other urogenital, breast, gynaecological and, soft tissue sarcomas and melanomas; patients with a new diagnosis of metastatic disease will be also included;
* Eligible for active treatment;
* Written informed consent to participate in the study.

Exclusion Criteria:

* Impossibility to undertake the expected measurements;
* Impossibility to guarantee the attendance of the follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed adult cancer patients, candidate for active treatment consecutively identified in 12 Italian IRCCS members of the ACC WG "Survivorship Care e Supporto Nutrizionale". Identification of consecutive cancer patients can be done over two weeks a month only, for the centres with the higher patients' load.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Percentage of patients who are alive.

SECONDARY OUTCOMES:
Progression-free survival | 1 year and 2 years
  Percentage of patients who are free from tumor progression.
Treatment toxicity | 1 year
  Treatment-related severe adverse event (grade > or =3) according to Common Terminology Criteria for Adverse Events (CTCAE v5.0) and toxicity resulting in any treatment delay or dose reduction.

CONTACTS AND LOCATIONS:
Locations (16):
- Italy (16):
  - IRCCS Istituto Tumori Giovanni Paolo II,, Bari, BA
  - IRCCS Saverio De Bellis, Castellana Grotte, BA
  - Istituto Ortopedico Rizzoli, Bologna, BO
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" IRCCS, Meldola, FC
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - IRCCS Ospedale San Raffaele, Milano, Milan, MI
  - Centro di Riferimento Oncologico, Aviano, PN
  - IOV Istituto Oncologico Veneto, Padua, PV
  - AUSL IRCCS Reggio-Emilia, Reggio Emilia, RE
  - IDI IRCCS - Istituto Dermopatico dell'Immacolata, Roma, RM
  - Istituto Nazionale Tumori Regina Elena, Roma, RM
  - Policlinico Universitario Agostino Gemelli, Roma, RM
  - Istituto di Candiolo - Fondazione del Piemonte per l'Oncologia - IRCCS, Candiolo, TO
  - IRCCS Sacro Cuore Don Calabria, Negrar, VR
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia

IPD SHARING:
Plan to Share IPD: Undecided
Data derived from the study are property of the Promoter, who will commit to sharing them with the Investigators of each participating centres and to publish the results of the study in order to give full and timely information to the scientific community. The results of the research could be communicated to third parties and made public in conferences by the Investigators after accordance with the Study Responsible, in compliance with the Ministerial Decree of 2.05.2006.

REFERENCES:
- [Background] Caccialanza R, De Lorenzo F, Gianotti L, Zagonel V, Gavazzi C, Farina G, Cotogni P, Cinieri S, Cereda E, Marchetti P, Nardi M, Iannelli E, Santangelo C, Traclo F, Pinto C, Pedrazzoli P. Nutritional support for cancer patients: still a neglected right? Support Care Cancer. 2017 Oct;25(10):3001-3004. doi: 10.1007/s00520-017-3826-1. Epub 2017 Jul 14. No abstract available. PMID 28710645
- [Background] Caccialanza R, Goldwasser F, Marschal O, Ottery F, Schiefke I, Tilleul P, Zalcman G, Pedrazzoli P. Unmet needs in clinical nutrition in oncology: a multinational analysis of real-world evidence. Ther Adv Med Oncol. 2020 Feb 14;12:1758835919899852. doi: 10.1177/1758835919899852. eCollection 2020. PMID 32110247
- [Background] Pedrazzoli P, Caccialanza R, Cotogni P, Degli Esposti L, Perrone V, Sangiorgi D, Di Costanzo F, Gavazzi C, Santoro A, Pinto C. The Advantages of Clinical Nutrition Use in Oncologic Patients in Italy: Real World Insights. Healthcare (Basel). 2020 May 6;8(2):125. doi: 10.3390/healthcare8020125. PMID 32384639